CLINICAL TRIAL: NCT03788369
Title: Evaluation of Effectiveness and Safety of Hybrid Coronary Revascularization, a Non-randomized, Prospective, Open-label Registry in Real-world Practice
Brief Title: Evaluation of Effectiveness and Safety of Hybrid Coronary Revascularization
Acronym: HCR registry
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2018-12
Record Dates: First submitted 2018-12-21; First posted 2018-12-27 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Percutaneous Coronary Revascularization; Coronary Stenosis; Coronary Artery Disease Progression; Coronary Artery Bypass Grafting
Keywords: Hybrid coronary revascularization
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multivessel coronary artery disease: must include left anterior descending artery
  Interventions: Procedure: Hybrid Coronary Revascularization

INTERVENTIONS:
Procedure: Hybrid Coronary Revascularization — Hybrid coronary revascularization (HCR) combines minimally invasive surgical coronary artery bypass grafting of the left anterior descending artery with percutaneous coronary intervention (PCI) of non-left anterior descending vessels.
  Other Names: HCR

SUMMARY:
This study evaluated the effectiveness and safety of Hybrid Coronary Revascularization in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 and more
* Hybrid coronary revascularization due to multivessel coronary artery disease(must include left anterior descending artery)
* Written consent

Exclusion Criteria:

* Previous CABG(coronary artery bypass graft)
* Life expectancy ≤1 year

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hybrid coronary revascularization due to multivessel coronary artery disease(must include left anterior descending artery)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
a composite event of death, myocardial infarction, TVR(Target Vessel Revascularization), or stroke. | 5 years
  Patients who have experienced any one of the following events are considered to have experienced the composite outcome: death, myocardial infarction, TVR(Target Vessel Revascularization), or stroke.

SECONDARY OUTCOMES:
All death | 5 years
Cardiac death | 5 years
Myocardial infarction | 5 years
a composite event of all death or myocardial infarction | 5 years
a composite event of cardiac death or myocardial infarction | 5 years
TVR(Target Vessel Revascularization) | 5 years
TLR(Target Lesion Revascularization) | 5 years
Stent thrombosis | 5 years
  by an Academic Research Consortium (ARC) category
Cerebrovascular event | 5 years
Procedural success | 5 days
  Procedural success is defined as < 30% final stenosis and the absence of in-hospital event including death, Q-wave myocardial infarction or urgent repeat revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided